CLINICAL TRIAL: NCT05770102
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations. Treatment Arm 02: Atezolizumab in Adult, Paediatric and Teenage/Young Adult Patients With Cancers With High TMB or MSI-high or Proven CMMRD Disposition.
Brief Title: DETERMINE Trial Treatment Arm 02: Atezolizumab in Adult, Paediatric and Teenage/Young Adult Patients With Cancers With High Tumour Mutational Burden (TMB) or Microsatellite Instability-high (MSI-high) or Proven Constitutional Mismatch Repair Deficiency (CMMRD) Disposition
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Manchester (Other); University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004 - Treatment Arm 2; IRAS ID: 1004057 (Other: IRAS)
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Malignancy; Malignant Neoplasm; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms by Site; Cancer; Colorectal Neoplasms; Endometrial Neoplasms; Melanoma; Solid Tumours
Keywords: Adult; Antineoplastic Agents; Atezolizumab; Cancer; Child; Malignancy; Malignant Neoplasms; Molecular Targeted Therapy; Neoplasms by Histologic Type; Neoplasms by Site; Paediatric; Precision Medicine; Rare; Tumour-agnostic; Young adult
MeSH Terms: conditions — Neoplasms; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms by Site; Colorectal Neoplasms; Endometrial Neoplasms; Melanoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 02: Atezolizumab (Experimental): This atezolizumab treatment arm is for adult, paediatric and TYA patients with cancers with high TMB or high MSI or proven (previously diagnosed) CMMRD.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Adult patients will receive 1200 mg of atezolizumab intravenously every 21 days.
  Paediatric patients will receive atezolizumab at a dose of 15 mg/kg (maximum 1200 mg) every 21 days.
  Patients may continue on treatment until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Tecentriq

SUMMARY:
This clinical trial is looking at a drug called atezolizumab. Atezolizumab is approved as standard of care treatment for adult patients with urothelial cancer, non-small cell lung cancer, extensive-stage small cell lung cancer, hepatocellular carcinoma and triple negative breast cancer. This means it has gone through clinical trials and been approved by the Medicines and Healthcare products Regulatory Agency (MHRA) in the UK.

Atezolizumab works in patients with these types of cancers which have certain changes in the cancer cells called high tumour mutational burden (TMB) or high microsatellite instability (MSI) or proven (previously diagnosed) constitutional mismatch repair deficiency (CMMRD).

Investigators now wish to find out if it will be useful in treating patients with other cancer types which are also TMB/MSH-high or show CMMRD. If the results are positive, the study team will work with the NHS and the Cancer Drugs Fund to see if these drugs can be routinely accessed for patients in the future.

This trial is part of a trial programme called DETERMINE. The programme will also look at other anti-cancer drugs in the same way, through matching the drug to rare cancer types or ones with specific mutations.

DETAILED DESCRIPTION:
DETERMINE Treatment Arm 02 (atezolizumab) aims to evaluate the efficacy of atezolizumab in adult, paediatric and teenage/young adult (TYA) patients with rare* cancers with high TMB or high MSI or proven CMMRD disposition and in common cancers where high TMB/MSI or proven CMMRD is considered to be infrequent.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients (includes paediatric and teenagers/young adult cancers) or common cancers with rare alterations.

This treatment arm has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

The ultimate aim is to translate positive clinical findings to the NHS (Cancer Drugs Fund) to provide new treatment options for rare adult, paediatric and TYA cancers.

OUTLINE:

Pre-screening: The Molecular Tumour Board (MTB) makes a treatment recommendation for the participant based on molecularly-defined cohorts.

Screening: Consenting patients undergo biopsy and collection of blood samples for research purposes.

Treatment: Patients will receive atezolizumab until disease progression without clinical benefit, unacceptable adverse events (AEs) or withdrawal of consent. Patients will also undergo collection of blood samples at various intervals while receiving treatment and at EoT.

After completion of study treatment, patients are followed up every 3 months for 2 years.

THE DETERMINE TRIAL MASTER (SCREENING) PROTOCOL:

Please see DETERMINE Trial Master (Screening) Protocol record (NCT05722886) for information on the DETERMINE Trial Master Protocol and applicable documents.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA WITHIN THE DETERMINE MASTER PROTOCOL (NCT05722886) AND WITHIN THE TREATMENT ARM 02 (ATEZOLIZUMAB) OUTLINED BELOW*

*When atezolizumab-specific inclusion/exclusion criteria or precautions below differ from those specified in the Master Protocol, the atezolizumab-specific criteria will take precedence.

Inclusion Criteria:

A. Confirmed diagnosis of a malignancy that is high TMB (defined as ≥10 mut/Mb), MSI-high or of proven (previously diagnosed) CMMRD disposition using an analytically validated next-generation sequencing method. Patient cases with TMB between 10-15 mut/Mb may be discussed in an MTB meeting. TMB ≥19 mut/Mb will be fast-tracked for an MTB recommendation, unless there are any patient-specific individualities (such as multiple gene amplifications) that require MTB discussion.

B. Women of childbearing potential are eligible provide they meet the following criteria:

* Have a negative serum or urine pregnancy test before enrolment and;
* Agree to use one form of effective birth control method such as:

I. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation ([oral, intravaginal or transdermal]);

II. progestogen-only hormonal contraception associated with or without inhibition of ovulation (oral, injectable or implantable);

III. intrauterine device (IUD),

IV. intrauterine hormone-releasing system (IUS),

V. bilateral tubal occlusion,

VI. vasectomised partner,

VII. sexual abstinence,

VIII. male or female condom with or without spermicide;

IX. cap, diaphragm or sponge with spermicide.

Effective from the first administration of atezolizumab, throughout the trial and for five months after the last administration of atezolizumab.

C. Male patients with partners who are women of childbearing potential are eligible provided that they agree to the following, from the first administration of atezolizumab, throughout the trial until the last administration of atezolizumab:

* Agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or sexual abstinence.
* Non-vasectomised male patients with partners who are women of childbearing potential must also be willing to ensure that their partner uses an effective method of contraception.
* Male patients with pregnant or lactating partners must be advised to use barrier method contraception (e.g. condom) to prevent drug exposure of the foetus or neonate.

All male patients must refrain from donating sperm for the same period.

D. Patients must be able and willing to undergo a fresh tissue biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow aspiration and/or trephine or lymph node biopsy samples may be taken.

E. ADULT PATIENTS (≥18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

F. PAEDIATRIC PATIENTS (<18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

G. Patients must have stable thyroid function tests. Patients on stable doses of thyroxine replacement are permitted.

Exclusion Criteria:

A. Diagnosis of urothelial cancer, non-small cell lung cancer, extensive-stage small cell lung cancer, hepatocellular carcinoma or triple negative breast cancer.

B. Patients with rapidly progressing or symptomatically deteriorating brain metastases and/or leptomeningeal disease. Patients with previously treated brain metastases are eligible, provided the patient has not experienced a seizure or had a clinically significant change in neurological status within 14 days (for adult patients) or 7 days (for paediatric patients) prior to the start of IMP administration. Such patients must be non-dependent on steroids or on a stable or reducing dose of steroid treatment for at least 14 days (or 7 days for paediatric patients) prior to the start of IMP administration. Primary brain or central nervous system (CNS) malignancies are allowed providing the patient is clinically stable (if requiring corticosteroids must be at stable or decreasing doses for at least 14 days for adults and 7 days for paediatric patients prior to the start of IMP administration). Patients who have received brain irradiation must have completed whole-brain radiotherapy and/or stereotactic radiosurgery at least 14 days prior to the start of IMP administration.

• Paediatric patients with either primary brain tumours or extracranial solid tumours with intracranial metastases with one or more intracranial lesions should only be considered for inclusion if largest intracranial lesion is ≤6 cm in longest axis. Consideration should also be given to the intracranial location of the tumour and potential risk should swelling occur. This is because of the class risk of immune checkpoint inhibitors such as atezolizumab causing immune-mediated inflammatory response and 'tumour flare' which may result in acute neurological deterioration.

C. Female patients who are pregnant, breastfeeding or planning to become pregnant during the trial or within five months following their last dose of atezolizumab.

D. History or clinical evidence of current inflammatory lung disease:

* History of idiopathic pulmonary fibrosis, organising pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* Evidence of active pneumonitis on screening chest computed tomography (CT) scan.

E. Active autoimmune disease that requires the use of systemic immunomodulatory therapy (i.e. with disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy for hypothyroidism and adrenal or pituitary insufficiency is acceptable.

F. Ongoing lung pathologies which, in the opinion of the Investigator present a compromise to safety (e.g. active tuberculosis).

G. Systemic immunomodulatory agents within 14 days prior to trial entry (immunostimulatory agents within four weeks). Exceptions to this are:

* Patients who received acute, low dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g. 48 hours of corticosteroids for a contrast allergy) are eligible for the trial.
* Patients who received corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma equivalent to ≤10 mg prednisolone a day or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the trial.
* Patients with primary CNS disease can be receiving concurrent treatment with corticosteroids. Patients must be receiving a stable or decreasing dose for ≥14 days for adults and ≥7 days for paediatric patients prior to the screening magnetic resonance imaging (MRI) scan and at the time of drug initiation.
* Patients who receive physiological doses of steroid replacement (e.g. hydrocortisone) are permitted.

H. Known to be serologically positive (as detected by polymerase chain reaction) for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).

I. History of severe allergic anaphylactic reactions to chimeric, human or humanised antibodies, or fusion proteins including other immune checkpoint inhibitors.

J. Known hypersensitivity to Chinese hamster ovary cell products.

K. Known hypersensitivity to atezolizumab or any of the excipients.

L. Patients who were administered a live, attenuated vaccine within 28 days prior to enrolment, or anticipation of need for such a vaccine during atezolizumab treatment or within six months after the final dose of atezolizumab.

M. Patients with clinically significant pre-existing cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or NYHA class III or IV congestive heart failure.

Patients with a cerebrovascular event (including stroke or transient ischaemic attacks [TIA]) or cardiovascular event (including acute myocardial infarction [MI]) within three months before the first dose of atezolizumab.

• Patients with primary CNS tumours may be considered unless intra-tumoural bleeding has occurred within 2 weeks of the first dose of atezolizumab, and patients with punctate CNS haemorrhages <3 mm may be considered.

Patients with a prior history of pericardial disorders, including pericarditis, pericardial effusion and cardiac tamponade.

N. Prior allogeneic stem cell or solid organ transplantation on immunosuppression.

O. Prior treatment with the same class of drug unless genetic profile demonstrates a mechanism of resistance known to be potentially sensitive to atezolizumab.

P. Uncontrolled diabetes.

Q. Any clinically significant concomitant disease or condition (or its treatment) that could interfere with the conduct of the trial or absorption of oral medications or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this trial.

R. Severe infection within four weeks prior to the first IMP administration or the administration of antibiotics within two weeks prior to the first IMP administration, with the exemption of patients requiring prophylaxis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  An OR is defined as the confirmed occurrence of either a Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 criteria (or immune related [ir]-RECIST or standard imaging criteria for specific disease e.g. Response Evaluation in Neuro Oncology criteria [RANO]). In patients with leukaemia, OR will be defined as the occurrence of CR, CRi (CR incomplete neutrophil recovery) or CRp (CR with incomplete platelet recovery). The trial will report the proportion of patients with an OR and 95% credible interval.
Durable Clinical Benefit (DCB) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  DCB is defined as the absence of disease progression for at least 24 weeks from the start of trial treatment according to RECIST Version 1.1 criteria (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) and, where relevant (e.g. for haematological malignancies), by standard bone marrow response assessment criteria. Alternative definitions of DCB based on different time points may be pre-specified for particular sub-cohorts if 24 weeks is not clinically relevant. The trial will report the proportion of patients with a DCB and 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DR) | Disease assessment every 2 cycles of atezolizumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of atezolizumab for up to 2 years.
  DR is defined as the time from the date of the first confirmed CR or PR according to RECIST 1.1 or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria to the date of disease progression. The trial will report the median DR and 95% credible interval.
Best percentage change in sum of target lesion / index lesion diameters (PCSD) | Disease assessment every 2 cycles of atezolizumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of atezolizumab for up to 2 years.
  PCSD is defined as the greatest decrease or least increase in the sum of target lesion diameters (RECIST) or index lesion diameters (irRECIST) as a percentage compared to the baseline measurement. The trial will report the mean PCSD and 95% credible interval.
Time to treatment discontinuation (TTD) | From first dose of atezolizumab to discontinuation of trial treatment up to 5 years.
  TTD is defined as the time from date of starting trial treatment to date of discontinuing trial treatment, in days estimated by the median of the posterior inverse gamma probability distribution. The trial will report the median TTD and 95% credible interval.
Progression-Free Survival time (PFS) | Disease assessment every 2 cycles of atezolizumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of atezolizumab for up to 2 years.
  PFS is defined as the time from date of starting trial treatment to date of progression or date of death without a previous progression recorded estimated by the median of the posterior inverse gamma probability distribution.
Time to Progression (TTP) | Disease assessment every 2 cycles of atezolizumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of atezolizumab for up to 2 years.
  TTP is defined as the time from date of starting trial treatment to date of progression or date of death without recorded progression censored rather than events. The trial will report the median TTP and 95% credible interval.
Growth Modulation Index (GMI) | Disease assessment every 2 cycles of atezolizumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of atezolizumab for up to 2 years.
  GMI is defined as the ratio of TTP with the trial protocol treatment to TTP on the most recent prior line of therapy. The trial will report the mean GMI and 95% credible interval.
Overall Survival time (OS) | Time of death or up to 2 years after the EoT visit.
  OS is defined as the time from date of starting trial treatment to date of death from any cause estimated by the median of the posterior normal probability distribution.
Occurrence of at least one Suspected Unexpected Serious Adverse Reaction (SUSAR) | From the time of consent until 90 days after last dose of atezolizumab (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  The trial will report the number of patients who experience at least one SUSAR to atezolizumab.
Occurrence of at least one Grade 3, 4 or 5 atezolizumab related AE | From the time of consent until 90 days after last dose of atezolizumab (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  Number of patients who experience at least one atezolizumab related Grade 3, 4 or 5 AE according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.
EORTC-QLQ-C30 Standardised Area Under Summary Score Curve (QLQSAUC) in adult patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For adult populations, multiple measures of Quality of Life (QoL) will be generated from patient completion of the European Organisation for Research and Treatment of Cancer QLQ-C30 (EORTC-QLQ-C30) questionnaire (15 measures). For each patient the Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean QLQSAUC and 95% credible interval.
EQ-5D Standardised Area Under Index Value Curve (EQ5DSAUC) in adult patients. | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For adult populations, two measures of QoL will be generated from patient completion of the EQ-5D-5L questionnaire. For each measure, scores based on responses from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean EQ5DSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in paediatric patients. | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For paediatric populations multiple measures of QoL will be generated from patient completion of the PedsQL 4.0 (4 measures). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in parents of paediatric patients. | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For paediatric populations multiple measures of QoL will be generated from patient's parent completion of the PedsQL 4.0 (4 measures). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (27):
- United Kingdom (27):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cardiff Children's Hospital, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Royal Hospital for Children Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Hospital, Liverpool
  - University College London Hospital, London
  - Guy's Hospital, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Great North Children's Hospital, Newcastle
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Sheffield's Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests for data relating to this treatment arm that are made within 5 years from last patient last visit for the atezolizumab treatment arm will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk

REFERENCES:
- See also: Overview of the DETERMINE trial. — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Master Screening Protocol (NCT05722886). — https://clinicaltrials.gov/ct2/show/NCT05722886